CLINICAL TRIAL: NCT00123123
Title: Oral Health and Ventilator-associated Pneumonia
Brief Title: Effect of Improved Oral Hygiene to Prevent Pneumonia in Hospitalized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Frank Scannapieco, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NIDCR-14685; R01DE014685 (NIH); 1R01-DE-14685-1A2
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2010-08

CONDITIONS: Pneumonia
Keywords: Ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Vehicle Control) (Placebo Comparator): Delivered Twice a day
  Interventions: Drug: placebo
- 0.12% chlorhexidine gluconate oral rinse (Experimental): Delivered twice a day
  Interventions: Drug: chlorhexidine gluconate oral rinse (0.12%)
- 0.12% chlorhexidine oral rinse (Experimental): Delivered once a day, placebo once a day
  Interventions: Drug: chlorhexidine gluconate oral rinse (0.12%); Drug: placebo

INTERVENTIONS:
Drug: chlorhexidine gluconate oral rinse (0.12%) — chlorhexidine gluconate oral rinse
  Arms: 0.12% chlorhexidine gluconate oral rinse; 0.12% chlorhexidine oral rinse
Drug: placebo
  Arms: 0.12% chlorhexidine oral rinse; Placebo (Vehicle Control)

SUMMARY:
Recent studies have found that poor oral hygiene may foster the colonization of the oropharynx by potential respiratory pathogens in mechanically-ventilated (MV), intensive care unit (ICU) patients. Thus, improvements in oral hygiene in MV-ICU patients may prevent ventilator-associated pneumonia (VAP).

The specific aims of this investigation are: 1) to organize the necessary infrastructure to develop and perform a pilot clinical trial to evaluate alternative oral hygiene procedures to prevent VAP; 2) to use this organization to perform a pilot clinical trial to determine if the use of oral topical chlorhexidine gluconate (CHX) will prevent dental plaque, oropharyngeal colonization by respiratory pathogens, and VAP in MV-ICU patients.

DETAILED DESCRIPTION:
Recent studies have found that poor oral hygiene may foster the colonization of the oropharynx by potential respiratory pathogens in mechanically-ventilated (MV), intensive care unit (ICU) patients. Thus, improvements in oral hygiene in MV-ICU patients may prevent ventilator-associated pneumonia (VAP). The Specific Aims of this investigation are: 1) to organize the necessary infrastructure to develop and perform a pilot clinical trial to evaluate alternative oral hygiene procedures to prevent VAP; 2) to use this organization to perform a pilot clinical trial to determine if the use of oral topical chlorhexidine gluconate (CHX) will prevent dental plaque, oropharyngeal colonization by respiratory pathogens, and VAP in MV-ICU patients. This pilot longitudinal, double blind intervention study will consider the appropriate frequency of delivery of CHX to improve oral hygiene in MV-ICU patients. Preliminary data from these pilot studies will also allow accurate sample size calculations to be made for a large-scale multi-center clinical trial; and 3) to perform molecular epidemiological studies to identify and genetically type bacteria cultured from lower airway secretions of MV-ICU patients with or without VAP and compare them to isolates of the same species from their dental plaque.

This pilot study will enable this multidisciplinary team of investigators to organize the infrastructure, patient recruitment and methodologic protocols, and data management and analysis procedures necessary to perform a multi-center, controlled clinical trial to assess the efficacy and generalizability of this intervention to improve oral hygiene in MV-ICU and prevent VAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study will be those admitted to the trauma intensive care unit (TICU) of Erie County Medical Center (ECMC) hospital. All patients admitted to the TICU who are intubated and mechanically ventilated within 24-48 hours of admission will be eligible for study admission, with the exception of those demonstrating the following exclusion criteria: a) a witnessed aspiration (to eliminate patients with chemical pneumonitis); b) a confirmed diagnosis of post-obstructive pneumonia (e.g. advanced lung cancer); c) a known hypersensitivity to CHX; d) patients for whom consent can not be obtained; e) a diagnosed thrombocytopenia (platelet count less than 40 and/or a INR above 2) or other coagulopathy; f) a do not intubate order; g) children under the age of 18 years; h) Pregnant women; i) Legal incarceration; j) If transferred from another ICU; k) Those with oral mucositis; l) Those with immunosuppression (either-HIV or drug induced [e.g. organ transplant patients or those on long term steroid therapy]); m) Patients re-admitted to the TICU
* Comatose and intubated patients will be included since they represent patients at greatest risk for respiratory infection.

Exclusion Criteria:

* Patients for whom consent can not be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Scannapieco, DMD PhD, Study Chair — University at Buffalo, The State University of New York; Frank A. Scannapieco, DMD PhD, Principal Investigator — The State University of New York
Locations (1):
- University of Buffalo, The State University of New York, Buffalo, New York, United States

REFERENCES:
- [Result] Scannapieco FA, Yu J, Raghavendran K, Vacanti A, Owens SI, Wood K, Mylotte JM. A randomized trial of chlorhexidine gluconate on oral bacterial pathogens in mechanically ventilated patients. Crit Care. 2009;13(4):R117. doi: 10.1186/cc7967. Epub 2009 Jul 15. PMID 19765321
- [Result] Heo SM, Haase EM, Lesse AJ, Gill SR, Scannapieco FA. Genetic relationships between respiratory pathogens isolated from dental plaque and bronchoalveolar lavage fluid from patients in the intensive care unit undergoing mechanical ventilation. Clin Infect Dis. 2008 Dec 15;47(12):1562-70. doi: 10.1086/593193. PMID 18991508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 March, 2004 until 30 November, 2007. Subjects were recruited from patients admitted to the ICU of the Erie County Medical Center (ECMC) who were mechanically ventilated. This ICU provides trauma, burn care, and rehabilitation and is an affiliated teaching facility for the State University of New York at Buffalo.
Groups:
- Placebo: Vehicle control twice a day (oral rinse)
- Chlorhexidine/Placebo: Chlorhexidine oral rinse 1 oz once a day/placebo oral rinse once a day
- Chlorhexidine: chlorhexidine 1 oz oral rinse twice a day
Period: Overall Study
Arm/Group | Placebo | Chlorhexidine/Placebo | Chlorhexidine
Started | 59 | 58 | 58
Completed | 59 | 58 | 58
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Chlorhexidine/Placebo | Chlorhexidine | Total
Number analyzed (Participants) | 59 | 58 | 58 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 59 | 58 | 58 | 175
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (22.5) | 44.8 (19.9) | 47.6 (19.1) | 48.0 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 14 | 52
  Male | 36 | 43 | 44 | 123
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 58 | 175

OUTCOME MEASURES:

1. Primary Outcome: Colonization of the Oral Cavity by Respiratory Pathogens (on Teeth/Denture/Buccal Mucosa) as Determined by Quantitative Cultures Expressed as Colony Forming Units (Cfu) Per ml (CFU/mL) of the Aerobic Cultivable Flora After 48 Hours
Description: Samples were diluted and plated on sheep's blood agar (to isolate S. aureus), and MacConkey agar (for isolation of Gram-negative bacilli) and incubated for 72 hours at 37°C in 5% carbon dioxide. Plates were assessed for growth for the following target bacteria: S. aureus, P. aeruginosa, Acinetobacter species, and enteric organisms (Klebsiella pneumoniae, Serratia marcescens, Enterobacter species, Proteus mirabilis, Escherichia coli). Results of quantitative cultures were expressed as colony forming units (cfu) per ml of sample.
Time Frame: Every 48 hours until discharge
Population: All tests were carried out using intent-to-treat analysis, with two-sided tests with a significance level of 0.05. Baseline comparisons between groups were made by analysis of variance (ANOVA) and/or the chi-squared test, as appropriate.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Placebo | Chlorhexidine/Placebo | Chlorhexidine
Number analyzed (Participants) | 59 | 58 | 58
CFU/mL | 7 (2) | 7.1 (1.9) | 5.1 (2)
Statistical Analysis 1: Comparison: Placebo vs Chlorhexidine/Placebo vs Chlorhexidine; A mixed effect model was used to compare overall treatment effects between groups for repeated measures data. The group comparison for each time point was performed using ANOVA; Test type: Superiority or Other; p = 0.6750, ANOVA

2. Secondary Outcome: Clinical Pulmonary Infection Score (CPIS) at 48 Hours
Description: The CPIS score was calculated as follows: 1) Fever: 0 (36.5 to 38.4°C), 1 (38.5 to 39), 2 (<36.0 OR >39.0); 2) Leukocytosis: 0 (4000 to 11,000 white blood cells per mm3 of blood), 1 (11,000 to 17,000), 2 (>17,000); 3) New infiltrate:
  0 = None, 1 = Patchy, 2 = Localized; 4) Secretions: 0 = None to minimal, 1 = moderate, 2 = large amount; and 5) PaO2/ FiO2: 0 = more than 330 and 2 = less than 330. Total scores for the subscales can range from 0-10, with lower scores indicating better outcome.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Chlorhexidine/Placebo | Chlorhexidine
Number analyzed (Participants) | 59 | 58 | 58
units on a scale | 2.5 (1) | 2.5 (0.9) | 2.4 (1)

ADVERSE EVENTS:
Time Frame: Patients were followed until discharge from the intensive care unit
Description: The numbers of participants at risk do not match numbers of participants provided in the participant flow module since some patients exited study before 48 hour assessment point.
Arm/Group | Placebo | Chlorhexidine/Placebo | Chlorhexidine
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/47 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No